CLINICAL TRIAL: NCT03759496
Title: Intravesical Administration of Durvalumab (MEDI4736) to Patients With High-risk, Non-muscle-invasive Bladder Cancer (NMIBC). A Phase II Study With Correlative
Brief Title: Efficacy of Durvalumab in Non-muscle-invasive Bladder Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hellenic GenitoUrinary Cancer Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-16-12611; 2018-002100-13 (EudraCT Number)
Record Dates: First submitted 2018-11-26; First posted 2018-11-30 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Bladder Cancer
Keywords: bladder; durvalumab; cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplasms | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab treated patients (Experimental): Subjects will receive up to 1000mg durvalumab (MEDI4736) via weekly intravesical administration, for up to a maximum of 6 weeks or until confirmed progression, unacceptable toxicity, withdrawal of consent, or another discontinuation criterion is met.
  Interventions: Biological: Durvalumab

INTERVENTIONS:
Biological: Durvalumab — Durvalumab is a human monoclonal antibody (mAb) of the immunoglobulin G (IgG) 1 kappa subclass
  Other Names: MEDI4736

SUMMARY:
Research Hypothesis Approximately 75% of patients with bladder cancer (BC) present with a disease confined to the mucosa (stage Ta, CIS) or submucosa (stage T1) (non-muscle invasive BC [NMIBC]). For high grade NMIBC, i.e. TaG3, T1G3 and CIS, intravesical bacillus Calmette-Guérin (BCG) immunotherapy is the treatment of choice, given that it prevents recurrence and reduces the odds of progression to MIBC. However, since initial BCG therapy fails in approximately 40% of patients over a 2-year period, new treatment options for these patients are of utmost importance.

In that field of research durvalumab, a human monoclonal antibody that binds programmed cell death ligand-1 (PD-L1), demonstrated meaningful clinical activity as well as manageable safety profile in PD-L1-positive patients with BC, many of whom were heavily pretreated. Certain studies using systemic administration of anti-PD1 agents for BCG refractory NMIBC are ongoing. Nevertheless, intravesical administration may be advantageous, since selective bladder tumor uptake of monoclonal antibodies following intravesical administration, while this method results in negligible absorption in the circulation and, therefore, minimal risk of systemic toxicity. This notion is supported by the findings of a recent study of intravesical administration of recombinant adenovirus-mediated interferon-α2b gene therapy (rAd-IFNα), No rAd-IFNα DNA was detected in the blood. Furthermore, no systemic toxicity was reported in a phase II study using the same agent.

The investigators, therefore, propose a phase II study of intravesical administration of durvalumab in patients with BCG refractory NMIBC. Since no safety or efficacy data specifically on intravesical administration of durvalumab exist, a run-in part will precede the main phase II, in order to confirm safety of the procedure and to reject a futility hypothesis, as described in the following sections of the protocol. Correlative studies of potential biomarkers in tumor tissue before and after durvalumab instillation are also proposed.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and any locally-required authorization (eg, HIPAA in the USA, EU Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
2. Age > 18 years at time of study entry
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Body weight >30kg
5. Diagnosis of high grade, non-muscle invasive urothelial carcinoma. High-grade carcinoma includes the following types

   1. TaG3
   2. T1G3
   3. CIS
6. Tumors with combinations of the above types or containing low grade components in addition to the high-grade component are acceptable. Disease refractory to Bacillus Calmette Guerin (BCG) therapy to adequate BCG exposure. BCG refractory disease is defined as

   1. If high-grade tumor appears during BCG therapy
   2. If high-grade, non-muscle-invasive papillary tumor is present at three months
   3. If CIS (with or without concomitant papillary tumor) is present at three and six months Adequate exposure is defined as a minimum of 5 out of 6 BCG induction doses. Μaintenance or re-induction can be used according to local practice but are not mandatory for the definition of adequate exposure.
7. High grade recurrence after an initial response to BCG therapy.
8. Patients intolerant to adequate BCG exposure, defined as

   1. fewer than 5 instillations of BCG induction therapy
   2. No more than one cycle of maintenance BCG therapy
9. Subjects may have received other intravesical or systemic therapies XML File Identifier: goagJWHcccRmyt+fBE00IC1ok+0= Page 12/26 for NMIBC or CIS before or after receiving BCG, as long as they meet the aforementioned criteria for BCG refractory disease.
10. Subjects are not candidates for immediate cystectomy or have elected not to undergo the procedure.
11. Adequate normal organ and marrow function as defined below:

    1. Haemoglobin ≥ 9.0 g/dL
    2. Absolute neutrophil count (ANC) > 1500 per mm3
    3. Platelet count >100,000 per mm3
    4. Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
    5. AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 5x ULN
    6. Serum creatinine Cl>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance
12. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal subjects. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    1. Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
    2. Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
13. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up

Exclusion Criteria:

1. Disease of the upper urinary tract or prostatic urethra
2. ECG with QTcF value >470 ms
3. Participation in another clinical study with an investigational product during the last 4 weeks
4. Concurrent enrolment in another clinical study, unless it is an observational (non interventional) clinical study or during the follow-up period of an interventional study
5. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) within 14 days prior to the first dose of study drug. Immediate postoperative intravesical instillation of epirubicin or mitomycin C is allowed if occurred more than 14 days prior to the first dose of the study drug.
6. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria Subjects with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician. Subjects with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
7. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer related conditions (eg, hormone replacement therapy) is acceptable.
8. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
9. History of allogenic organ transplantation.
10. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]) - more details in protocol.
11. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
12. History of another primary malignancy with exceptions described in protocol
13. History of leptomeningeal carcinomatosis
14. History of active primary immunodeficiency
15. Active infection including tuberculosis, hepatitis B, hepatitis C, or human immunodeficiency virus. Subjects with a past or resolved HBV infection are eligible. Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA (see details in protocol)
16. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab with exceptions described in protocol
17. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Subjects, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
18. Female subjects who are pregnant or breastfeeding or male or female subjects of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
19. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
20. Prior randomization or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) of Durvalumab among 500mg, 750mg and 1000mg that will be given intravesically to patients with BCG-refractory NMIBC | 6 months after trial initiation
The possibility of a rate of high-grade relapse free (HGFR) that it is defined as the development of TaG3, T1G3, CIS or muscle-invasive disease after the initiation of durvalumab therapy. | 6 months after trial initiation
Efficacy of intravesical administration of Durvalumab at MTD in patients with BCG-refractory NMIBC assessed by 1-year high-grade-relapse-free (HGRF)-rate | 1 year after patient enrollment

SECONDARY OUTCOMES:
Toxicity of the MTD of intravesical Durvalumab administration assessed according to the NCI CTC version 4.03 except from local irritation. | 6 months after trial initiation
  Local irritation will be assessed according to the following criteria: Grade 1: Microscopic hematuria Grade 2: Moderate frequency. Intermittent macroscopic hematuria. Grade 3: Severe frequency and dysuria. Frequent hematuria. Reduction in bladder capacity (<150 cc) Grade 4: Necrosis/ Contracted bladder (capacity <100 cc). Severe hemorrhagic cystitis
Efficacy assessed by the high-grade progression-free rate at 30 days after the last durvalumab instillation and 6 months following durvalumab therapy. | 30 days and 6 month after last durvalumab instillation
PD-L1 and VEGF expression assessed in tumor tissue obtained before and after durvalumab instillation | 33 months after FPFV
  Immunohistochemistry will be used for the evaluation of PD-L1 and VEGF expression levels
Assessment of PD-L1 and VEGF protein levels in urine samples obtained before and after durvalumab instillation | 33 months after FPFV

CONTACTS AND LOCATIONS:
Locations (1):
- Hellenic GenitoUrinary Cancer Group, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fragkoulis C, Bamias A, Gavalas N, Tzannis K, Fragiadis E, Pinitas A, Stamatakos PV, Papadopoulos G, Stathouros G, Grammatoglou X, Korkolopoulou P, Zoubouli C, Stravodimos K, Ntoumas K, Mitropoulos D, Skolarikos A, Papatsoris A. Intravesical Administration of Durvalumab for High-risk Non-muscle-invasive Bladder Cancer: A Phase 2 Study by the Hellenic GU Cancer Group. Eur Urol. 2025 Mar;87(3):281-284. doi: 10.1016/j.eururo.2024.12.018. Epub 2025 Jan 17. PMID 39827021